CLINICAL TRIAL: NCT02541396
Title: A Pilot Study Of The Efficacy Of WafermineTM Alone And In Combination With Opioids In Subjects Undergoing Bunionectomy
Brief Title: A Study Of The Effectiveness Of Wafermine Alone And In Combination With Opioids In Subjects Undergoing Bunionectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: iX Biopharma Ltd. (Other)
Collaborators: Jean Brown Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KET009
Record Dates: First submitted 2015-08-26; First posted 2015-09-04 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Acute Pain
Keywords: Bunion; Bunionectomy
MeSH Terms: conditions — Acute Pain; Bunion | interventions — Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Group A (Placebo Comparator): Placebo wafers given every 2 hours Placebo capsule given every 4 hours Placebo wafers "top-up" dose given at hour 1
  Interventions: Drug: Placebo
- Group B (Active Comparator): Placebo wafers given every 2 hours Oxycodone given every 4 hours Placebo wafers "top-up" dose given at hour 1
  Interventions: Drug: Oxycodone
- Group C (Experimental): Wafermine™ 35 mg wafer + placebo wafer given every 2 hours Placebo capsule given every 4 hours Wafermine™ 35 mg wafer + placebo wafer "top-up" dose at hour 1
  Interventions: Drug: Wafermine
- Group D (Experimental): Wafermine™ 35 mg wafer + placebo wafer given every 2 hours Oxycodone 5 mg capsule every 4 hours Wafermine™ 35 mg "wafer + placebo wafer top-up" dose at hour 1
  Interventions: Drug: Wafermine; Drug: Oxycodone
- Group E (Experimental): Wafermine™ 35 mg + placebo wafer given every 4 hours Placebo wafers given every 2 hours Placebo capsule given every 4 hours Wafermine™ 35 mg wafer + placebo wafer "top-up" dose at hour 1
  Interventions: Drug: Wafermine
- Group F (Experimental): Wafermine™ 35 mg + placebo wafer given every 4 hours Placebo wafers given every 2 hours Oxycodone 5 mg given every 4 hours Wafermine™ 35 mg wafer + placebo wafer "top-up" dose at hour 1
  Interventions: Drug: Wafermine; Drug: Oxycodone
- Group G (Experimental): Wafermine™ 70 mg given every 4 hours Placebo wafer given every 2 hours Placebo capsule given every 4 hours 2 Placebo wafers "top-up" dose at hour 1
  Interventions: Drug: Wafermine

INTERVENTIONS:
Drug: Wafermine — 35 or 70 mg ketamine in a sublingual wafer
  Other Names: Sublingual ketamine
  Arms: Group C; Group D; Group E; Group F; Group G
Drug: Oxycodone — 5 mg oxycodone capsule
  Arms: Group B; Group D; Group F
Drug: Placebo — Placebo capsule or placebo wafer
  Arms: Group A

SUMMARY:
To evaluate the safety and effectiveness of Wafermine administered with and without an opioid medication for acute pain following bunionectomy surgery.

DETAILED DESCRIPTION:
This is a Phase 2, randomised, double-blind, double-dummy, placebo-controlled evaluation of the analgesic efficacy and safety of WafermineTM alone and in combination with low-dose oxycodone in adult subjects who experience post-operative pain after undergoing primary unilateral bunionectomy. The study will randomise sufficient subjects to have 72 completed subjects at 1 site.

Study subjects will receive multiple doses of study medication over a 14 hour period and will be asked to complete pain and relief assessments as well as tolerability questionnaires over a 24 hour period.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for a bunionectomy (with no additional procedures).
* Healthy, ambulatory subjects able to understand and willing to comply with study procedures, study restrictions and requirements.
* Body mass index (BMI) ≥19 to ≤33 kg/m2.
* Females: Not pregnant, not lactating, and not planning to become pregnant during the study.
* Females: Be abstinent, surgically sterile, at least two years post-menopausal; or medically acceptable contraception.
* Able to read and understand English.
* Able to swallow oral capsules whole.

Exclusion Criteria:

* Allergy, intolerance, or contraindication to ketamine, oxycodone, morphine, ibuprofen or surgical medications.
* Clinically significant medical condition.
* History of illicit drug use or alcohol abuse and not in full remission.
* Positive test for human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) at the screening visit.
* Clinically significant 12 lead ECG abnormalities at screening.
* Smokers who are unwilling to abstain during the inpatient stay.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Total Pain Relief (TOTPAR) | 24 hours
  Subjects will use an 11 point numerical pain rating scale (NPRS) where 0=No Pain and 10= Worst Possible pain to rate their pain at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, 11.5, 12, 12.5, 13, 13.5, 14, 14.5, 15, 15.5, 16 and 24 hours.
  TOTPAR is computed as follows at the specified time points: TOTPAR-t = ∑ [T(i) - T(i-1) * [(PR(i-1) + PR(i))/2]

SECONDARY OUTCOMES:
Percent with maximum Pain Relief | 24 hours
  The percent of maximum pain relief is defined as the proportion of subjects reporting "Complete Relief" (score of 4) on a 4 point categorical scale (no relief, a little relief, some relief, a lot of relief and complete relief) at each time point over the sampling interval.
Proportion of Subjects requiring "Rescue Medication" | 24 hours
  Calculation of the proportion of subjects requiring "Rescue Medication" at each time point over the sampling interval.
Time to onset of perceptible and meaningful pain relief | 24 hours
  Calculated using the double stopwatch technique. Subjects stop the first stopwatch when they experience perceptible relief and the second stopwatch when they experience meaningful relief.
Time to onset of complete pain relief (Peak Relief) | 24 hours
  Measurement of the time it takes subjects to report their maximum pain relief on a 5 point categorical relief scale (0=no relief, 1=a little relief, 2=some relief, 3=a lot of relief, 4=complete relief)
Time to maximum reduction in pain intensity | 24 hours
  Measurement of the time it takes subjects to reach their maximum reduction in pain on the 11 point NPRS where 0=No pain and 10=Worst Possible pain.
Time for pain intensity to return to baseline | 24 hours
  Measurement of the time for pain intensity to return to baseline using scores from the NPRS assessments where 0=No pain and 10=Worst possible pain.
Time to rescue medication | 24 hours
  Measurement of the time elapsed from initial dose of study medication to time of first dose of rescue medication.
Percentage of Maximum Total Pain Relief (TOTPAR) | 24 hours
  Subjects will use an 11 point numerical pain rating scale (NPRS) where 0=No Pain and 10= Worst Possible pain to rate their pain at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, 11.5, 12, 12.5, 13, 13.5, 14, 14.5, 15, 15.5, 16 and 24 hours. Percentage of Maximum Total Pain Relief is computed at each time-point using:
  %maxTOTPAR= 〖TOTPAR〗_t/〖maxTOTPAR〗_t x100
Sum of Pain Intensity Differences (SPID) | 24 hours
  Subjects will use an 11 point numerical pain rating scale (NPRS) where 0-No Pain and 10= Worst Possible pain to rate their pain at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, 11.5, 12, 12.5, 13, 13.5, 14, 14.5, 15, 15.5, 16 and 24 hours.
  Sum of Pain Intensity Differences is computed at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 8.5, 9, 9.5, 10, 10.5, 11, 11.5, 12, 12.5, 13, 13.5, 14, 14.5, 15, 15.5, 16 and 24 hours. SPIDx is a time weighted sum of pain intensity difference score from baseline over the time interval in hours.
Responder Rates (30% and 50%) | 24 hours
  The responder rate is defined as the proportion of subjects with a value of percentage change greater than or equal to 30% (and 50%) from baseline in pain intensity (using scores from the 11 point NPRS where 0=no pain and 10=worst possible pain) at each time point over the sampling interval.
Safety (treatment emergent adverse events, significant changes in physical examination findings as well as vital sign measurements) | 24 hours
  Measurement of treatment emergent adverse events reported during the study. Measurement of significant changes in physical examination findings as well as vital sign measurements (heart rate, blood pressure, breathing rate and pulse oximetry readings).
Tolerability (judged by subject answers on oral symptoms questionnaire) | 24 hours
  Measurement of tolerability as judged by subject answers on oral symptoms questionnaire measuring irritation, burning and bitterness, as well as physical examination of oral cavity. Also measuring the number of subjects who discontinue the study due to intolerable side effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Jean Brown Research, Salt Lake City, Utah, United States